CLINICAL TRIAL: NCT04377022
Title: Effect of Aerobic Exercise Training on Balance, Walking Capacity, and Quality of Life in Sub-acute Stroke.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Ishtiaq Ahmed, Physiotherapist, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 342
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Cerebrovascular Stroke; Cerebrovascular Accident, Acute; Cerebral Stroke
Keywords: Aerobic exercise; Stroke; Walking Capacity
MeSH Terms: conditions — Stroke | interventions — Psychotherapy, Multiple; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Therapy (No Intervention): In this group, Patients receive Conventional Therapy for 40 minutes daily and 5 days in a week. The training period was 5 week after the recruitment of patients.
- Combined Therapy (Experimental): In this group, Patients receive Aerobic exercise training in addition to conventional Physical Therapy. Patients undergoes Aerobic exercise training for 25 minutes and 3 days in a week. A total of 15 session of aerobic exercise training session was given to patient.
  Interventions: Other: Combined Therapy (Aerobic Exercise in addition to conventional therapy)

INTERVENTIONS:
Other: Combined Therapy (Aerobic Exercise in addition to conventional therapy) — There are two intervention arm in the study
  1. Combined therapy
  2. Conventional Therapy
  Arms: Combined Therapy

SUMMARY:
Stroke is one of the major cause of morbidity and mortality and the leading cause of disability in adults all around the world. Stroke survivors can suffer several neurological impairments and deficits which have an important impact on patient's quality of life and which increase the costs for health and social services. After stroke, impairments in ADLs and functional status, deterioration in health related quality of life can be seen.

The purpose of this study is to Determine the effect of Aerobic exercise training on Balance, Walking capacity and quality of life in sub-acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age.
* Stroke that occurred in the recent 3 months.
* Who can walk independently or by using assistive device.
* Have a minimum Chedoke McMaster Stroke Assessment (CMSA) leg impairment score of 3 but less than 7.

Exclusion Criteria:

* Patients were excluded from the study if they have a stroke that occurs more than 3 months.
* If resting blood pressure more than 160/100 even after taking medications
* Have by-pass surgery in recent 3 months.
* Other musculoskeletal problems which restrict the patient's ability to do aerobic activity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
6 Minute walk Test: | 5 week
  To measure the physical performance of individual after stroke.

SECONDARY OUTCOMES:
Berg Balance test and rating scale | 5 week
  It is use o measure the Balance and stability of patient. Total score of the scale is 56. A score of < 45 indicates individuals may be at greater risk of falling.
Stroke Impact scale | 5 week
  To measure the impairment and quality of life after stroke. The maximum score is 140.

CONTACTS AND LOCATIONS:
Overall Officials: Awais bin Inam, MSOMPT, Principal Investigator — Government College University, Faislabad
Locations (1):
- Bin-Inam Rehabilitation Clinic Faisalabad, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No